CLINICAL TRIAL: NCT01933906
Title: Phase 1 Study to Evaluate the Feasibility and Efficacy of the Addition of P1101 (PEG-Proline-Interferon Alpha-2b) to Imatinib Treatment in Patients With Chronic Phase Chronic Myeloid Leukaemia Not Achieving a Complete Molecular Response (MR 4.5 or BCR-ABL Transcripts Not Detectable)
Brief Title: Addition of P1101 to Imatinib Treatment in Patients With Chronic Phase Chronic Myeloid Leukaemia Not Achieving a Complete Molecular Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_CML 1; 2013-000115-24 (EudraCT Number)
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
Keywords: CML; Chronic myeloid leukemia; Chronic myeloid leukaemia; PEG-Proline-Interferon-alpha 2b; Interferon; P1101; Imatinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1101 (Experimental): P1101 50µg s.c. will be administered every 2 weeks in addition to preexisting imatinib treatment. In the absence of dose limiting toxicities after 12 weeks, the dose will be escalated to 100µg every 2 weeks.
  Maximum treatment duration will not expand 18 months.
  Interventions: Drug: P1101

INTERVENTIONS:
Drug: P1101
  Other Names: PEG-Proline-Interferon alpha-2b

SUMMARY:
In this phase I pilot study, it is planned to investigate the feasibility and safety of adding an interferon therapy to an preexisting imatinib treatment in patients with chronic phase chronic myeloid leukaemia. The participating patients have already reached a response during their imatinib therapy (CCyR) but have still a detectable disease (no molecular response MR 4.5 or better).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* BCR-ABL positive chronic myeloid leukaemia in chronic phase treated with imatinib as first line therapy
* CHR, CCyR after at least 18 months of imatinib treatment
* Adequate organ function, defined as the following:

  * total bilirubin < 1.5 x ULN,
  * AST and ALT < 2.5 x ULN,
  * creatinine < 1.5 x ULN,
  * ANC > 1.5 x 109/L,
  * platelets > 100 x 109/L
* Written, voluntarily signed informed consent

Exclusion Criteria:

* CMR (molecular remission 4.5 or BCR-ABL transcripts undetectable)
* Patient has received any other investigational treatment within 28 days before study entry
* Treatment with a second generation tyrosine kinase inhibitor (dasatinib, nilotinib)
* ECOG performance status ≥ 3
* Patients with a primary of a different histological origin than the study indication (unless relapse-free interval is ≥ 5 years, except cervical carcinoma, basal cell epithelioma or squamous cell carcinoma of the skin)
* Evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease etc.)
* Acute chronic infections
* Known autoimmune disease (e.g. collagen disease, polyarthritis, immune thrombocytopenia, thyroiditis, psoriasis, lupus nephritis or any other autoimmune disorder)
* Female patients who are pregnant or breast-feeding
* Known diagnosis of HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Number and seriousness of adverse events to evaluate safety and tolerability | 30 months
  The primary objective is to determine the safety and tolerability of the addition of P1101 to the pre-study established dose of imatinib.

SECONDARY OUTCOMES:
Efficacy (Number of patients achieving an improvement of remission status) | 30 months
  Secondary objective is to determine the rate of achievement of ≥ 1 log reduction from the initial BCR-ABL transcript level at study entry and the achievement of molecular remission 4.5 or undetectable BCR-ABL transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Thaler, MD, Study Director — Klinikum Wels-Grieskirchen GmbH
Locations (4):
- Austria (4):
  - Klinikum Wels-Grieskirchen GmbH, IV. Interne Abteilung, Wels, Upper Austria
  - Universitätskliniken Innsbruck, Univ.-Klinik f.Innere Medizin V Hämtologie u. Onkologie, Innsbruck
  - Ordensklinikum Linz - Elisabethinen, Linz
  - Universitätsklinikum der PMU Salzburg, Universitätsklinik für Innere Medizin III, Salzburg

IPD SHARING:
Plan to Share IPD: No